CLINICAL TRIAL: NCT04238026
Title: Distal Radial Artery Approach to Prevent Radial Artery Occlusion
Brief Title: Distal Radial Artery Approach to Prevent Radial Artery Occlusion (DAPRAO)
Acronym: DAPRAO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Responsible Party: Principal Investigator, Joaquin Jimenez-Castellanos, MD, Instituto Nacional de Cardiologia Ignacio Chavez
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: INCAR-DG-DI-386-2019
Record Dates: First submitted 2020-01-18; First posted 2020-01-23 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Radial Artery Occlusion
MeSH Terms: conditions — Arterial Occlusive Diseases

STUDY DESIGN:
Intervention Model Description: Two randomized groups, one receiving traditional radial access and the other receiven distal radial access
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Distal radial artery approach (Experimental): Puncture in the snuff box area of the arm with through and through technique, advancement of a wire and placement of an hydrophilic sheath introducer.
  Interventions: Procedure: Distal radial artery approach
- Proximal radial artery approach (Active Comparator): Puncture in the ventral side of the arm (2 cm proximal to the styloid apophysis) with through and through technique, advancement of a wire and placement of an hydrophilic sheath introducer.
  Interventions: Procedure: Distal radial artery approach

INTERVENTIONS:
Procedure: Distal radial artery approach — Use of distal radial artery approach in coronary angiography and angioplasty

SUMMARY:
The main complication of transradial intervention is radial artery occlusion (RAO). This is relevant because it limits the radial approach for future interventions and disables this conduit for coronary bypass grafts and arteriovenous fistula. Observational studies suggest that distal radial access could reduce RAO incidence.

The primary endpoint of our study is to compare the efficacy of the distal and proximal transradial approaches in terms of RAO incidence. The safety endpoint is the incidence of complications between these two methods.

ELIGIBILITY:
Inclusion Criteria:

* Perceptible radial artery pulse
* Diagnostic or interventional procedure feasible to be performed with radial access.

Exclusion Criteria:

* Myocardial infarction with ST segment elevation in time for primary angioplasty.
* Cardiogenic shock or hemodynamic instability.
* Clinical, plethysmography or ultrasound suggestive of occlusion of the radial artery
* Prior recent radial artery access (1 month)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of our study is to compare the efficacy of the distal and proximal transradial approaches in terms of RAO incidence. | The RAO will be evaluated 24 hours after the procedure by ultrasound examination and was defined as the absence of both color pattern and pulsed wave registry.
  The primary endpoint of our study is to compare the efficacy of the distal and proximal transradial approaches in terms of RAO incidence.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Cardiology, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes